CLINICAL TRIAL: NCT03046199
Title: Detection of COPD in Primary Care
Acronym: DISCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 35RC16_9770_DISCO
Record Dates: First submitted 2017-02-01; First posted 2017-02-08 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention)
- Questionnaire (Experimental)
  Interventions: Other: Questionnaire
- Coordination (Experimental)
  Interventions: Other: Coordination
- Questionnaire + coordination (Experimental)
  Interventions: Other: Questionnaire; Other: Coordination

INTERVENTIONS:
Other: Questionnaire — Targeted screening of COPD by GPs via the GOLD / HAS questionnaire. The questionnaire includes 4 questions for patients over 40. At least one positive response is an indication to perform a spirometry.
  Arms: Questionnaire; Questionnaire + coordination
Other: Coordination — Information of the GPs of the existence of a coordination of the care of proximity to facilitate the access to the spirometry (identification of a referent specialist, making appointments).
  Arms: Coordination; Questionnaire + coordination

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common chronic disease with a significant medical and economic impact. Its prevalence is increasing and is estimated at 7.5% of people over 40 in France. COPD is responsible for a significant impairment of quality of life and was the 3rd leading cause of death in the world in 2010 when it was 4th place 20 years ago.

However, about 75% of patients with COPD are not diagnosed. Spirometry is the only examination for the diagnosis of COPD. Patients identified at risk for COPD are insufficiently using spirometry and general practitioners (GPs) underestimate the severity of COPD when they do not practice spirometry in their patients. COPD is often diagnosed too late, the disease being discovered at the stage of complications requiring hospitalization. The underdiagnosis is mainly due to poor knowledge of patients, their difficulty in accessing a specialist performing spirometry, their reluctance to perform spirometry, and the insufficient involvement of general practitioners.

Currently in France, targeted screening for COPD and diagnosis in primary care is a major challenge. The international (GOLD 2014) and French (HAS 2014) recommendations do not indicate a systematic screening in the general population for COPD but advocate targeted screening of patients by five questions to identify risk factors and symptoms of COPD. The presence of at least one of these factors in an adult over the age of 40 requires spirometry.

Recent studies suggest the relevance of finding primary care variables for smoking and respiratory symptoms in order to identify new cases of COPD.

However, the impact of the use of these questionnaires on the prevalence of diagnoses of COPD in general practice has not been demonstrated. Moreover, the heterogeneity of the provision of care according to the territories limits a fast or easy access (distance) to the spirometry.

It is therefore necessary to evaluate in primary care the interest of a targeted screening of COPD and the interest of a coordination of care for the realization of a spirometry, in order to improve the rate of diagnosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with health insurance
* Non-opposition to participation in the study

Exclusion Criteria:

* COPD known and confirmed by spirometry
* Asthma known and confirmed by spirometry
* Patient not having the physical or mental ability to perform spirometry
* Pregnant woman
* Patient under protection
* Patient already included in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3162 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of COPD in each of the study's 4 arms, to assess the relevance of each intervention and the interaction between these interventions. | 6 months
  Prevalence is defined as the number of patients with positive spirometry (i.e FEV1 / post-bronchodilator CVF <0.70) in relation to the number of patients included.

SECONDARY OUTCOMES:
Distribution of the severity stages of COPD | 6 months
  Severity stage will be evaluated with FEV1 in each arm
Time to diagnosis of COPD according to the GOLD / HAS score | 6 months
Prevalence of COPD according to the GOLD / HAS score | 6 months
Severity of COPD according to the GOLD / HAS score | 6 months
Time to spirometry | 6 months
  Delay between consultation with GP and realization of a spirometry when applicable in each arm
Number of spirometries performed in each arm | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chapron A, Pele F, Andres E, Fiquet L, Laforest C, Veislinger A, Fougerou C, Turmel V, Fouchard J, Yourish B, Oumari S, Allory E, Banatre A, Schweyer FX, Pommier J, Brinchault G, Guillot S, Laviolle B, Jouneau S. [Targeted screening of COPD in primary care: Feasibility and effectiveness]. Rev Mal Respir. 2019 Feb;36(2):162-170. doi: 10.1016/j.rmr.2018.08.023. Epub 2019 Jan 24. French. PMID 30686560